CLINICAL TRIAL: NCT05685303
Title: Safety and Efficacy of the Alleviant System for No-Implant Interatrial Shunt Creation in Patients With Chronic Heart Failure
Brief Title: Alleviant ALLAY-HF Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Alleviant Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CIP-0003
Record Dates: First submitted 2022-12-14; First posted 2023-01-17 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Subjects randomized to the treatment arm will undergo cardiac imaging, femoral vein access and receive the Alleviant ALV1 System device procedure.
  Interventions: Device: Alleviant ALV1 System
- Control (Sham Comparator): Subjects randomized to the control arm will undergo cardiac imaging and sheath placement in femoral vein.
  Interventions: Other: Sham-Control

INTERVENTIONS:
Device: Alleviant ALV1 System — Creation of interatrial shunt
  Arms: Treatment
Other: Sham-Control — Cardiac imaging
  Arms: Control

SUMMARY:
Prospective, multicenter, randomized, sham-controlled, double blinded, adaptive study designed to evaluate the safety and efficacy of a percutaneously created interatrial shunt using the Alleviant ALV1 System in patients with HFpEF/HFmrEF.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic HFpEF/HFmrEF with LVEF greater than or equal to 40%
2. NYHA Class II, III or ambulatory IV
3. Exercise right heart catheterization*

   1. Elevated left atrial pressure during exercise right heart catheterization (greater than or equal to 25 mmHg)
   2. Exercise PVR < 1.8 WU
4. Ongoing stable GDMT

Exclusion Criteria:

1. Advanced heart failure
2. Presence of a pacemaker
3. Evidence of right heart dysfunction

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite Primary Endpoint | 12-month
  The primary endpoint is a composite of mortality, heart failure events and quality of life based on Kansas City Cardiomyopathy Questionnaire (KCCQ) calculated at 12 months. KCCQ responses are provided along a rating scale from 0-100 with a higher score indicating better health.

CONTACTS AND LOCATIONS:
Overall Officials: James Udelson, MD, Principal Investigator — Tufts Medical Center
Locations (90):
- United States (53):
  - University of Alabama, Birmingham, Alabama
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Pima Heart and Vascular, Tucson, Arizona
  - Memorial Care Long Beach Medical Center, Long Beach, California
  - UC Davis Medical Center, Sacramento, California
  - Scripps Clinical Research Services, San Diego, California
  - San Francisco VA, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Hartford Hospital, Hartford, Connecticut
  - The Cardiac and Vascular Institute (TCAVI), Gainesville, Florida
  - HCA Florida Memorial Hospital, Jacksonville, Florida
  - NCH Research Institute, Naples, Florida
  - Advent Health Orlando, Orlando, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Atlanta VA Health Care System, Decatur, Georgia
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins Medical Institution, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - VA Ann Arbor, Ann Arbor, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Washington University - St Louis, St Louis, Missouri
  - VA NY Harbor Healthcare System, New York, New York
  - New York University, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - South Oklahoma Heart Research, LLC., Oklahoma City, Oklahoma
  - Providence St. Vincent's Medical Center, Portland, Oregon
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - Prisma Health - Midlands, Columbia, South Carolina
  - Monument Health, Rapid City, South Dakota
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Hendrick Health, Abilene, Texas
  - Austin Heart, Austin, Texas
  - UT Southwestern, Dallas, Texas
  - Baylor Scott & White Research Institute, Plano, Texas
  - NextStage Clinical Research, Waco, Texas
  - University of Washington, Seattle, Washington
  - Advocate Aurora Health/Aurora Research Institute, Milwaukee, Wisconsin
- Australia (2):
  - Monash Health Victorian Heart Hospital, Clayton, Victoria
  - Royal Adelaide Hospital, Adelaide
- Medizinische Universität Graz, Graz, Austria
- Belgium (3):
  - OLV Hospital, Aalst
  - ZNA Middelheim, Antwerp
  - AZ Sint Jan Brugge, Bruges
- Canada (3):
  - Southlake Regional Hospital Centre, Newmarket, Ontario
  - Centre hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Centre Integre Universitaire de Sainte et de Services Scoiiaux de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke (CIUSSS de l'Estrie - CHUS), Montreal, Quebec
- Tbilisi Heart and Vascular, Tbilisi, Georgia
- Germany (9):
  - Heart and Vascular Center-Bad Bevensen, Bad Bevensen
  - Herz- und Gefasszentrum Bad Bevensen, Bad Bevensen
  - University of Gießen, Giessen
  - Marienkrankenhaus, Hamburg
  - Askelepios Klinik Altona, Hamburg
  - St. Vincentius Kliniken, Karlsruhe
  - Universitatsklinikum Schleswig-Holstein (UKSH), Lübeck
  - Universitätsklinikum Kardiologie, Magdeburg
  - Universitatsmedizin Rostock, Rostock
- European Interbalken Medical Center, Thessaloniki, Greece
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Shamir Medical Center, Zrifin
- Italy (2):
  - Humanitas Research Milan, Rozzano, MI
  - Instituto Auxologico Italiano, Milan
- New Zealand (2):
  - ChristChurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- Poland (4):
  - Poznan University of Medical Sciences, Poznan
  - 4th Military Hospital, Wroclaw
  - Uniwesytecki Szpital Kliniczny, Wroclaw
  - Silesian Center for Heart Disease, Zabrze
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Barcelona Hospital del Mar, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Valencia Hospital Clinico, Valencia

IPD SHARING:
Plan to Share IPD: No